CLINICAL TRIAL: NCT00401375
Title: A Phase 3, Double-Blind, Randomized, Parallel-Group, Placebo-Controlled Study of Intravenous (IV) Methylnaltrexone Bromide (MNTX) in the Treatment of Post-Operative Ileus (POI)
Brief Title: Study of Intravenous (IV) Methylnaltrexone Bromide (MNTX) in the Treatment of Post-Operative Ileus (POI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MNTX 3301
Record Dates: First submitted 2006-11-16; First posted 2006-11-20 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Post-Operative Ileus (POI)
MeSH Terms: interventions — methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- MNTX 12 mg (Experimental): Participants will receive methylnaltrexone (MNTX) 12 milligrams (mg) as an intravenous (IV) infusion over approximately 20 minutes for every 6 hours until one of the following occurs: 1) 24 hours elapsed after the first bowel movement and the participant was tolerating clear liquids, 2) the participant was discharged from the hospital, or 3) a maximum of 10 days elapsed. The first dose of study drug will be administered within the first 90 minutes after the end of surgery (defined as the time when the last skin suture or staple is placed in the participant).
  Interventions: Drug: Methylnaltrexone
- MNTX 24 mg (Experimental): Participants will receive MNTX 24 mg as an IV infusion over approximately 20 minutes for every 6 hours until one of the following occurs: 1) 24 hours elapsed after the first bowel movement and the participant was tolerating clear liquids, 2) the participant was discharged from the hospital, or 3) a maximum of 10 days elapsed. The first dose of study drug will be administered within the first 90 minutes after the end of surgery (defined as the time when the last skin suture or staple is placed in the participant).
  Interventions: Drug: Methylnaltrexone
- Placebo (Placebo Comparator): Participants will receive placebo matching to MNTX as an IV infusion over approximately 20 minutes for every 6 hours until one of the following occurs: 1) 24 hours elapsed after the first bowel movement and the participant was tolerating clear liquids, 2) the participant was discharged from the hospital, or 3) a maximum of 10 days elapsed. The first dose of study drug will be administered within the first 90 minutes after the end of surgery (defined as the time when the last skin suture or staple is placed in the participant).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylnaltrexone — Methylnaltrexone will be administered as per the dose and schedule specified in the respective arms.
  Other Names: MNTX
  Arms: MNTX 12 mg; MNTX 24 mg
Drug: Placebo — Placebo matching to methylnaltrexone will be administered as per the schedule specified in the respective arm.
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of MNTX in participants who have undergone segmental colectomy and to assess if the time between the end of surgery and the first bowel movement is significantly shorter in the MNTX regimen than the equivalent assessment using a placebo regimen.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants at least 18 years of age.
* All participants must meet American Society of Anesthesiologists (ASA) physical status I, II, or III.
* Participants must sign an informed consent form (ICF).
* Participants must be scheduled for a segmental colectomy via open laparotomy with general anesthesia.
* Females of childbearing potential must have a negative serum pregnancy test at the screening visit.
* Negative for history of chronic active hepatitis B, hepatitis C or Human Immunodeficiency Virus (HIV) infection.

Exclusion Criteria:

* Participants who received any investigational new drug in the 30 days prior to screening visit.
* Females who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2006-10-31 (Actual); Primary Completion 2008-02-29 (Actual); Study Completion 2008-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Mathew, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Progenics Pharmaceuticals, Tarrytown, New York, United States

REFERENCES:
- [Derived] Yu CS, Chun HK, Stambler N, Carpenito J, Schulman S, Tzanis E, Randazzo B. Safety and efficacy of methylnaltrexone in shortening the duration of postoperative ileus following segmental colectomy: results of two randomized, placebo-controlled phase 3 trials. Dis Colon Rectum. 2011 May;54(5):570-8. doi: 10.1007/DCR.0b013e3182092bde. PMID 21471758
- See also: Related Info — http://www.progenics.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Postoperative participants (who underwent segmental colectomy via open laparotomy) were randomized in 1:1:1 ratio to MNTX 12 mg, MNTX 24 mg, or placebo treatment groups. Randomization was based on regional stratification.
Groups:
- MNTX 12 mg: Participants received methylnaltrexone (MNTX) 12 milligrams (mg) as an intravenous (IV) infusion over approximately 20 minutes for every 6 hours until one of the following occurred: 1) 24 hours elapsed after the first bowel movement and the participant was tolerating clear liquids, 2) the participant was discharged from the hospital, or 3) a maximum of 10 days elapsed. The first dose of study drug was administered within the first 90 minutes after the end of surgery (defined as the time when the last skin suture or staple was placed in the participant).
- MNTX 24 mg: Participants received MNTX 24 mg as an IV infusion over approximately 20 minutes for every 6 hours until one of the following occurred: 1) 24 hours elapsed after the first bowel movement and the participant was tolerating clear liquids, 2) the participant was discharged from the hospital, or 3) a maximum of 10 days elapsed. The first dose of study drug was administered within the first 90 minutes after the end of surgery (defined as the time when the last skin suture or staple was placed in the participant).
- Placebo: Participants received placebo matched to MNTX as an IV infusion over approximately 20 minutes for every 6 hours until one of the following occurred: 1) 24 hours elapsed after the first bowel movement and the participant was tolerating clear liquids, 2) the participant was discharged from the hospital, or 3) a maximum of 10 days elapsed. The first dose of study drug was administered within the first 90 minutes after the end of surgery (defined as the time when the last skin suture or staple was placed in the participant).
Period: Overall Study
Arm/Group | MNTX 12 mg | MNTX 24 mg | Placebo
Started | 174 | 176 | 174
Received at Least 1 Dose of Study Drug (Modified intent-to-treat (mITT)/Safety population) | 171 | 173 | 171
Completed | 152 | 151 | 149
Not Completed | 22 | 25 | 25
Not completed — Protocol Violation | 2 | 2 | 1
Not completed — Adverse Event | 6 | 11 | 10
Not completed — Withdrawal by Subject | 9 | 7 | 7
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Other than specified | 2 | 1 | 3
Not completed — Randomized but not treated | 3 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Groups:
- MNTX 12 mg: Participants received MNTX 12 mg as an IV infusion over approximately 20 minutes for every 6 hours until one of the following occurred: 1) 24 hours elapsed after the first bowel movement and the participant was tolerating clear liquids, 2) the participant was discharged from the hospital, or 3) a maximum of 10 days elapsed. The first dose of study drug was administered within the first 90 minutes after the end of surgery (defined as the time when the last skin suture or staple was placed in the participant).
- Total: Total of all reporting groups
Arm/Group | MNTX 12 mg | MNTX 24 mg | Placebo | Total
Number analyzed (Participants) | 171 | 173 | 171 | 515
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (15.5) | 58.2 (15.6) | 58.1 (15.6) | 57.7 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 71 | 77 | 227
  Male | 92 | 102 | 94 | 288

OUTCOME MEASURES:

1. Primary Outcome: Time to First Bowel Movement
Description: Time to first bowel movement was measured from the end of surgery (defined as the time when the last skin suture or staple was placed in the participant). Time of the first bowel movement was recorded on the electronic case report form (eCRF). The first bowel movement was defined as a normal stool for a postoperative participant based on the clinical judgment of the investigator or designee. Analysis was performed by Kaplan-Meier estimate. Participants who had a bowel movement but were readmitted to the hospital within 1 week after discharge with a diagnosis of postoperative ileus (POI) were considered censored at the time of the first bowel movement as if the bowel movement had not occurred.
Time Frame: Day 1 (From the time of end of surgery [that is; from the first dose of study drug administration]) up to Day 10
Population: mITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Error); unit: days
Arm/Group | MNTX 12 mg | MNTX 24 mg | Placebo
Number analyzed (Participants) | 171 | 173 | 171
days | 4.4 (0.13) | 4.8 (0.21) | 4.6 (0.15)
Statistical Analysis 1: Comparison: MNTX 24 mg vs Placebo; Treatment comparisons were made at the overall α=0.05 level (2-sided) using a closed sequential procedure. Placebo and MNTX 24 mg groups were compared first; Test type: Other; p = 0.4259, Log Rank — Threshold for significance at 0.05 level; Mean Difference (Final Values) = -0.23
Statistical Analysis 2: Comparison: MNTX 12 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.3575, Log Rank — Threshold for significance at 0.05 level; Mean Difference (Final Values) = 0.13

2. Secondary Outcome: Time to Discharge Eligibility
Description: Time to discharge eligibility was measured from the end of surgery (defined as the time when the last skin suture or staple was placed in the participant). Discharge eligibility was defined as both tolerance of solid food and at least one bowel movement. Participants were considered to have tolerated solid food when they have eaten greater than or equal to (≥) 50 percent (%), of the first of two successive solid food meals (based on the judgement of the investigator or designee), without vomiting or nausea. Participants readmitted to the hospital with a diagnosis of POI within 7 days of discharge were considered treatment failures. Analysis was performed by Kaplan-Meier estimate.
Time Frame: Day 1 (From the time of end of surgery [that is; from the first dose of study drug administration]) up to Day 10
Population: mITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Error); unit: days
Arm/Group | MNTX 12 mg | MNTX 24 mg | Placebo
Number analyzed (Participants) | 171 | 173 | 171
days | 5.8 (0.24) | 7.0 (0.45) | 6.5 (0.32)

3. Secondary Outcome: Time to Discharge Order Written From the End of Surgery
Description: The investigator or designee recorded the time of the order. Participants re-admitted to the hospital with a diagnosis of POI within 7 days after discharge were considered treatment failures. Analysis was performed by Kaplan-Meier estimate.
Time Frame: Day 1 (From the time of end of surgery [that is; from the first dose of study drug administration]) up to Day 10
Population: mITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Error); unit: days
Arm/Group | MNTX 12 mg | MNTX 24 mg | Placebo
Number analyzed (Participants) | 171 | 173 | 171
days | 6.8 (0.26) | 9.1 (0.76) | 7.3 (0.29)

4. Secondary Outcome: Number of Participants With Clinically Meaningful Events (CMEs) for Nausea or Retching/Vomiting at 0 or 24 Hours as Evaluated by the Opioid-Related Symptom Distress Scale (SDS)
Description: CMEs were defined using opioid-related SDS (assessed participant-reported levels of severity concerning 10 symptoms associated with opioid medication usage: fatigue, drowsiness, inability to concentrate, nausea, dizziness, constipation, itching, difficulty with urination, confusion and retching/vomiting). CME = any symptom rated as severe (3) or very severe (4), with the exception of confusion. A total CME score was calculated by summing the number of CMEs across symptoms and ranged from 0 to 9. CME was counted for either nausea or vomiting/retching, or both and reported in this outcome measure.
Time Frame: 0 and 24 hours
Population: mITT population included all randomized participants who received at least 1 dose of study drug. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | MNTX 12 mg | MNTX 24 mg | Placebo
Number analyzed (Participants) | 171 | 173 | 171
Participants
  Nausea | 13 | 12 | 17
  Vomiting/Retching | 9 | 4 | 5

ADVERSE EVENTS:
Time Frame: Day 1 (From the time of end of surgery [that is; from the first dose of study drug administration]) up to end of follow-up visit (Day 17)
Description: Safety population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | MNTX 12 mg | MNTX 24 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 26/171 | 33/173 | 38/171
Other Adverse Events (participants affected / at risk) | 121/171 | 124/173 | 138/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MNTX 12 mg (N=171) | MNTX 24 mg (N=173) | Placebo (N=171)
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Colonic stenosis (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatic fistula (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Peritoneal effusion (Gastrointestinal disorders) | 0 | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 3 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2 | 3
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 3 | 2
Abdominal infection (Infections and infestations) | 1 | 0 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 0 | 1
Incision site cellulitis (Infections and infestations) | 0 | 1 | 0
Incision site infection (Infections and infestations) | 1 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 1 | 0
Pelvic abscess (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 3 | 0
Postoperative wound infection (Infections and infestations) | 1 | 1 | 1
Sepsis (Infections and infestations) | 3 | 4 | 4
Septic shock (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 1 | 1 | 2
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 6 | 6 | 6
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Failure to anastomose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 2 | 0
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0 | 0
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 3 | 2 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 3 | 5
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 3 | 1 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 1 | 0
General nutrition disorder (Metabolism and nutrition disorders) | 0 | 0 | 1
Colon cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MNTX 12 mg (N=171) | MNTX 24 mg (N=173) | Placebo (N=171)
Anaemia (Blood and lymphatic system disorders) | 19 | 14 | 10
Tachycardia (Cardiac disorders) | 22 | 21 | 10
Abdominal distension (Gastrointestinal disorders) | 13 | 17 | 15
Abdominal pain (Gastrointestinal disorders) | 24 | 22 | 15
Constipation (Gastrointestinal disorders) | 9 | 11 | 10
Diarrhoea (Gastrointestinal disorders) | 12 | 7 | 14
Dyspepsia (Gastrointestinal disorders) | 6 | 9 | 7
Nausea (Gastrointestinal disorders) | 73 | 64 | 83
Vomiting (Gastrointestinal disorders) | 21 | 24 | 31
Pyrexia (General disorders) | 27 | 33 | 47
Urinary tract infection (Infections and infestations) | 10 | 4 | 11
Procedural hypotension (Injury, poisoning and procedural complications) | 9 | 8 | 9
Procedural pain (Injury, poisoning and procedural complications) | 30 | 25 | 28
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 10 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 21 | 20 | 26
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 13 | 3
Headache (Nervous system disorders) | 8 | 12 | 11
Anxiety (Psychiatric disorders) | 12 | 9 | 14
Insomnia (Psychiatric disorders) | 10 | 10 | 17
Dysuria (Renal and urinary disorders) | 2 | 3 | 9
Urinary retention (Renal and urinary disorders) | 7 | 11 | 13
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 12 | 7 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 10 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 19 | 22 | 19
Hypertension (Vascular disorders) | 19 | 22 | 16
Hypotension (Vascular disorders) | 16 | 18 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.